CLINICAL TRIAL: NCT03719430
Title: A Phase II Trial Evaluating APX005M (a CD40 Agonistic Monoclonal Antibody) in Combination With Standard-of-Care Doxorubicin for the Treatment of Advanced Sarcomas
Brief Title: APX005M and Doxorubicin in Advanced Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander Z. Wei, MD (Other)
Collaborators: Apexigen America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alexander Z. Wei, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS0095
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: Leiomyosarcoma; Liposarcoma; Pleomorphic sarcoma; Synovial sarcoma; Malignant peripheral nerve sheath tumor; Spindle cell sarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Neurofibrosarcoma | interventions — Doxorubicin; sotigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doxorubicin/APX005M (Experimental): Patients will be treated with doxorubicin and APX005M in 21 day cycles. All patients receive the same treatment (there is no "placebo" arm). After completing 8 cycles of study treatment, patients without evidence of disease progression or unacceptable toxicity may continue treatment with APX005M alone. Doxorubicin will not be continued beyond cycle 8 due to the risk for cardiac toxicity from cumulative dosing.
  Interventions: Drug: Doxorubicin; Drug: APX005M

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin is an anthracycline antibiotic with antineoplastic activity 75 mg/m2 IV day 1 (21 day cycles)
  Other Names: ADRIAMYCIN
Drug: APX005M — APX005M is a CD40 agonistic monoclonal antibody 0.3 mg/kg IV day 1 (21 day cycles)
  Other Names: APX-005M

SUMMARY:
This phase II clinical trial will evaluate the safety and efficacy of adding APX005M (a CD40 agonistic monoclonal antibody) to doxorubicin for the treatment of patients with advanced soft tissue sarcoma. The investigators believe that doxorubicin, which is currently the standard of care for most advanced sarcomas, could work better when combined with APX005M, which is a type of immunotherapy.

DETAILED DESCRIPTION:
Doxorubicin, a chemotherapy, is currently considered standard-of-care treatment for most advanced soft tissue sarcomas. This study will assess the safety and efficacy of combining APX005M, a novel immunomodulatory drug, together with standard of care doxorubicin, for the treatment of patients with advanced soft tissue sarcoma. APX005M is an agonistic monoclonal antibody targeting the CD40 receptor and may have favorable effects on certain types of immune cells in sarcoma tumors, particularly macrophages.

The primary objective is to determine the objective response rate. Secondary objectives include further evaluation of safety and efficacy. A subset of patients will undergo tumor biopsies at baseline and while on study treatment to help understand how the drug combination works and to evaluate how the composition of immune cells in the tumor changes after the treatment.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed advanced soft tissue sarcoma for which doxorubicin treatment is considered appropriate. Patients with well-differentiated liposarcoma who have histologic evidence of a dedifferentiated component are eligible. Kaposi sarcoma and gastrointestinal stromal tumor (GIST) are not eligible. Protocol Amendment 4 restricts further enrollment to participants with the following sarcoma subtypes. A total of 10 patients will be enrolled with each of the following sarcoma subtypes for the entire study, inclusive of patients enrolled prior to Amendment 4:

   * Dedifferentiated liposarcoma
   * Leiomyosarcoma
   * Myxofibrosarcoma/undifferentiated pleomorphic sarcoma
2. Disease must be locally advanced and unresectable or metastatic (that is, considered not amenable to curative surgery or radiation).
3. Patients must have measurable disease by RECIST criteria version 1.1.
4. Patients must demonstrate an ECOG performance status of 0 or 1 and be considered an appropriate candidate for anthracycline chemotherapy. There is no limit on prior lines of systemic therapy received. Treatment naïve patients may be enrolled.
5. Acceptable laboratory parameters:

   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥ 100,000/mm3
   * Creatinine ≤ 1.5 times upper limit of normal OR Calculated creatinine clearance > 45 mL/min
   * Total bilirubin ≤ upper limit of normal
   * AST/ALT ≤ 1.5 times upper limit of normal
6. Patients must have normal left ventricular systolic function, as demonstrated by a transthoracic echocardiogram or MUGA scan at screening, showing a normal left ventricular ejection fraction as defined by the laboratory performing the test.
7. Women of child-bearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of study drug administration.
8. Ability to understand and willingness to sign a written informed consent document.
9. After the safety lead-in phase is complete, the next consecutive 10 patients enrolled on the study must have a site of tumor tissue which is amenable to image-guided biopsy by interventional radiology with at most minimal risk to the patient. These 10 patients will be required to undergo tumor biopsy at screening and while on-treatment.

Exclusion Criteria

1. Patients must not have received treatment with any chemotherapy, immunotherapy, radiotherapy or an investigational agent for malignancy within the 21 days preceding registration. Patients may not have received treatment with a small molecule targeted anti-cancer agent within 14 days preceding study registration, provided this represents at least 7 half-lives for that agent. Furthermore, toxic effects from any prior therapy (except alopecia) must have resolved to ≤ grade 1 by NCI CTCAE v 5.0 or to the patient's baseline by registration.
2. Patients may not be receiving any other investigational agent for any purpose.
3. Patients may not have received prior treatment with:

   * any anthracycline chemotherapy
   * CD40 agonist
4. Patients may not have received prior radiotherapy of the mediastinal or pericardial area or whole pelvis radiation.
5. Patients may not have active, known or suspected autoimmune disease with the exceptions of well-controlled: asthma or allergic rhinitis, vitiligo, type 1 diabetes mellitus, psoriasis, or hypothyroidism.
6. Patients may not be receiving chronic systemic steroid therapy in excess of physiologic/ replacement doses (prednisone ≤ 10 mg/day is acceptable), or on any other form of immunosuppressive medication for 14 days prior to registration.
7. Patients with symptomatic brain metastases may not be enrolled. Those subjects with untreated brain metastases ≤ 1 cm who are asymptomatic and for whom there are no plans for surgery, radiation or corticosteroid use may be considered eligible at the discretion of the principal investigator. Subjects with brain metastases that have been treated and are stable for at least 30 days are eligible if asymptomatic and not receiving corticosteroids. Screening for brain metastases is not required and should not be routinely pursued given their uncommon incidence in sarcoma.
8. Patients may not have:

   * uncontrolled intercurrent illness including, but not limited to congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmias, uncontrolled diabetes mellitus or uncontrolled psychiatric illness that would limit compliance with study requirements in the opinion of the investigator.
   * unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction within 6 months of registration.
   * any thromboembolic event within 1 month prior to registration
   * any active coagulopathy
   * any clinically serious, active infection requiring treatment with antibiotics within 14 days prior to registration
   * major surgery within 28 days of registration.
9. Patients may not have history of another primary cancer, with the exception of:

   * curatively treated non-melanomatous skin cancer,
   * curatively treated cervical carcinoma in-situ,
   * other primary cancers treated with curative intent, no known active disease and no treatment administered within 2 years prior to registration.
   * other cancers considered indolent and for which no treatment is anticipated, in the opinion of the principal investigator
10. Patients may not be pregnant or nursing.
11. Patients may not have known HIV or hepatitis A, B or C infection; however, screening tests for these infections are not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  The percentage of patients achieving a partial or complete response as measured by imaging assessments from study treatment

SECONDARY OUTCOMES:
Recommended Dose Combination for APX005M and Doxorubicin and Combination Treatment | 6 months
  A safety-lead in phase will be conducted during which a small number of patients will be treated and monitored closely for certain side effects. If these side effects are seen, the dose of doxorubicin will be adjusted and the study treatment reassessed among another small number of patients. The purpose of the safety lead-in phase is to establish a safe and tolerable dose combination ("the recommended dose") which will be used during the remainder of the study.
Evaluation of Side Effects from APXO05M and Doxorubicin Treatment | 18 months
  Patients on the study will be assessed at regular intervals during clinical visits and through laboratory testing to monitor side effects from the study treatment.
Progression Free Survival | 18 months
  The mean time to either disease progression or death, whichever comes first, for patients on the study
Objective Response Rate (ORR) | 1 year
  Objective response rate in patients with dedifferentiated liposarcoma, leiomyosarcoma, and myxofibrosarcoma/undifferentiated pleomorphic sarcoma. The confirmed ORR per RECIST version 1.1. criteria will be evaluated in the group of patients with these 3 sarcoma subtypes and within each of these subtypes.

OTHER OUTCOMES:
Changes in Immune Cell Infiltrates in Baseline and On-Study Biopsies | 18 months
  Correlative/Exploratory Study
Expression of CD40 in Baseline Study Biopsies | 18 months
  Correlative/Exploratory Study

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wei, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Columbia University Irving Medical Center/NYP, New York, New York

IPD SHARING:
Plan to Share IPD: No